CLINICAL TRIAL: NCT06176079
Title: Pilot Study of Magnetic Resonance Imaging With Hyperpolarized Pyruvate (13C) In Patients With Fatty Liver Disease
Brief Title: Hyperpolarized Pyruvate (13C) Magnetic Resonance Imaging In Patients With Fatty Liver Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Michael Ohliger, MD PhD (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, Michael Ohliger, MD PhD, Principal Investigator, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Other Study IDs: 19-29381; 5R01DK115987 (NIH)
Record Dates: First submitted 2023-12-10; First posted 2023-12-19 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Non Alcoholic Fatty Liver; Non Alcoholic Steatohepatitis; NAFLD; NASH
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be obtained.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Part 1 (Cohort A): No injection of hyperpolarized (HP) 13C: Participants who are comprised of, primarily, healthy volunteers will undergo a standard MRI scan.
  Interventions: Procedure: Magnetic Resonance Imaging
- Part 1 (Cohort B): Injection of hyperpolarized (HP) 13C or HP13C-pyruvate+HP13C-urea "copol": Participants will receive HP 13C injection, and receive an MRI scan. Imaging results will be used to optimize the hyperpolarized 13C part of the imaging procedure. Participants will also have the option of undergoing repeated dose imaging studies of HP 13C-pyruvate or HP13C-pyruvate+HP13C-urea "copol", (up to a total of two injections per imaging visit separated by 15-60 minutes). Participants may be asked to fast up to 6 hours prior to the scan and the initial HP 13C MRI scan may be taken while participants are in a fasted state. Participants who have fasted will be offered up to 20 ounces (oz) of an oral glucose, fructose, or other high calorie drink (i.e. Gatorade, Coca-Cola, Ensure, etc.) to increase blood glucose levels, and a second HP 13C MRI scan will be performed after caloric intake.
  Interventions: Drug: Hyperpolarized (HP) 13C; Drug: Hyperpolarized 13C-Urea; Procedure: Magnetic Resonance Imaging; Procedure: Saline Flush
- Part 2 (Group 1): NAFLD: Participants with diagnosed NAFLD will receive HP 13C-pyruvate or HP13C-pyruvate+HP13C-urea "copol" injection optimized in Part 1 of the study as well as standard liver MRI pulse sequences.
  Interventions: Drug: Hyperpolarized (HP) 13C; Drug: Hyperpolarized 13C-Urea; Procedure: Magnetic Resonance Imaging; Procedure: Saline Flush
- Part 2 (Group 2): NASH: Participants with diagnosed NASH will receive HP 13C-pyruvate or HP13C-pyruvate+HP13C-urea "copol" injection optimized in Part 1 of the study as well as standard liver MRI pulse sequences.
  Interventions: Drug: Hyperpolarized (HP) 13C; Drug: Hyperpolarized 13C-Urea; Procedure: Magnetic Resonance Imaging; Procedure: Saline Flush
- Part 2 (Group 3): Healthy Volunteers: Healthy volunteers without known liver disease will receive HP 13C-pyruvate or HP13C-pyruvate+HP13C-urea "copol" injection optimized in Part 1 of the study as well as standard liver MRI pulse sequences.
  Interventions: Drug: Hyperpolarized (HP) 13C; Drug: Hyperpolarized 13C-Urea; Procedure: Magnetic Resonance Imaging; Procedure: Saline Flush

INTERVENTIONS:
Drug: Hyperpolarized (HP) 13C — A dosage of 0.43 mL/kg body weight at the maximum dosage will be injected intravenously at a rate of 5 mL/second.
  Other Names: HP 13C
  Groups: Part 1 (Cohort B): Injection of hyperpolarized (HP) 13C or HP13C-pyruvate+HP13C-urea "copol"; Part 2 (Group 1): NAFLD; Part 2 (Group 2): NASH; Part 2 (Group 3): Healthy Volunteers
Drug: Hyperpolarized 13C-Urea — Given intravenously (IV)
  Other Names: HP13C-urea; copol
  Groups: Part 1 (Cohort B): Injection of hyperpolarized (HP) 13C or HP13C-pyruvate+HP13C-urea "copol"; Part 2 (Group 1): NAFLD; Part 2 (Group 2): NASH; Part 2 (Group 3): Healthy Volunteers
Procedure: Magnetic Resonance Imaging — Imaging procedure
  Other Names: MRI; MR
Procedure: Saline Flush — A 20 milliliter (mL) saline flush at 5 mL/second will be given after each dose of HP 13C
  Groups: Part 1 (Cohort B): Injection of hyperpolarized (HP) 13C or HP13C-pyruvate+HP13C-urea "copol"; Part 2 (Group 1): NAFLD; Part 2 (Group 2): NASH; Part 2 (Group 3): Healthy Volunteers

SUMMARY:
The recent development of dissolution dynamic nuclear polarization (DNP) technology for hyperpolarized (HP) 13C imaging offers a promising new avenue for non-invasively accessing fundamental metabolic changes associated with the progression of fatty liver disease in vivo. The purpose of this pilot study is to optimize sequence parameters for hyperpolarized 13C acquisition in the human liver and determine which metabolic changes can be seen in humans with simple, non-alcoholic fatty liver disease (NAFLD) and non-alcoholic steatohepatitis (NASH) when compared to healthy volunteers.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

1. Optimize scan parameters in order to maximize the signal-to-noise ratio of the HP 13C-pyruvate magnetic resonance imaging (MRI) in the liver.
2. Determine whether the level of lactate production (as measured by the lactate/pyruvate ratio) in NASH participants, participants with simple NAFL, and healthy volunteers.

SECONDARY OBJECTIVES:

1. Develop data analysis methods to quantify HP C-13 pyruvate MRI data.
2. Further characterize the safety profile of HP C-13 pyruvate injections.

EXPLORATORY OBJECTIVES:

1. Examine the impact of the dual liver blood supply on the vascular kinetics of observed hyperpolarized 13C metabolism.
2. Improve methods of quantification and motion correction for hyperpolarized 13C acquisition, incorporating perfusion information derived from 13C Urea

OUTLINE:

Part 1: (Imaging Optimization, N=50): Participants enrolled in Part 1 will predominantly be healthy volunteers. As the protocol optimization is completed, there is a possibility that testing in using data from participants with fatty liver disease may be performed. Participants in this part will be divided into two cohorts:

* Cohort A: Participants will undergo MRI but no injection of hyperpolarized 13C.
* Cohort B: Participants will receive one HP 13C injection. Participants in this cohort will have the option of undergoing repeated dose imaging studies of HP 13C-pyruvate or HP 13C-pyruvate+HP 13C-urea "copol", for up to a total of two injections per imaging visit.

Part 2: (Pilot Study, N=30): Participants enrolled in Part 2 will receive the HP 13C-pyruvate or HP13C-pyruvate+HP13C-urea "copol" protocol that was optimized in Part 1 as well as standard liver MRI pulse sequences. Participants will be stratified into the following groups based on diagnosis:

* Group 1 (n=10): Participants with a diagnosis of non-alcoholic fatty liver without steatohepatitis (NAFL)
* Group 2 (n=10): Participants with a diagnosis of non-alcoholic steatohepatitis (NASH)
* Group 3 (n=10): Participants with no known liver disease (healthy volunteers)

Participants will be followed for 2-4 days following imaging procedure.

ELIGIBILITY:
Inclusion Criteria:

Part 1 (Imaging Optimization):

1. Able and willing to sign informed consent.
2. Age >= 18 years old at the time of study entry.

Part 2 (Pilot Study):

* Group 1 (Fatty Liver Patients without NASH):

  1. NAFL as determined by either clinical suspicion of fatty liver disease based on:

     1. steatosis by imaging or histology,
     2. no significant alcohol consumption,
     3. absence of coexisting liver disease OR NAFL determined by liver biopsy 3 months prior to the scan, with the presence of fat on histology but absent ballooning or fibrosis. (nonalcoholic steatohepatitis activity score (NAS) <= 3).
  2. Able and willing to sign informed consent.
  3. Age ≥ 18 years old at the time of study entry.
  4. Alcohol consumption < 2 drinks/day for men and <1 drink/day for women
  5. Hepatitis B surface antigen (HBsAg), Hepatitis C Virus (HCV) antibody, human immunodeficiency virus (HIV) antibody negative.
  6. Serum alanine aminotransferase (ALT) < 400 microliter (uL)
* Group 2 (NASH Patients):

  1. NASH as determined by liver biopsy 3 months prior to the scan.

     a) NASH defined as NAS score greater than or equal to 4 with confirmation of NASH by an anatomic pathologist.
  2. Able and willing to sign informed consent.
  3. Age >= 18 years old at the time of study entry.
  4. Alcohol consumption < 2 drinks/day for men and <1 drink/day for women
  5. HBsAg, HCV antibody, HIV antibody negative.
* Group 3 (Healthy volunteer):

  1. No known history of diabetes or liver disease.
  2. Able and willing to sign informed consent.
  3. Age >= 18 years old at the time of study entry.
  4. Body mass index < 25.
  5. Liver panel normal (aspartate aminotransferase (AST), ALT, alkaline phosphatase, bilirubin).
  6. HBsAg, HCV antibody, HIV antibody negative.
  7. Hemoglobin A1c < 5.7%.
  8. Estimated glomerular filtration rate (eGFR) >= 60 mL/min/1.73m^2

Exclusion Criteria:

Part 1 (Imaging Optimization): For Cohorts 1/B only:

1. Poorly controlled hypertension, with blood pressure at study entry > 160 mmHg systolic or > 100 mmHg diastolic.
2. Congestive heart failure with New York Heart Association (NYHA) status ≥ 2.
3. Pregnant or nursing.
4. Participants unwilling or unable to undergo magnetic resonance (MR) imaging, including participants with contra-indications to MRI, such as cardiac pacemakers or non-compatible intracranial vascular clips.
5. Participant size too large to fit in MR scanner.

Part 2 (Pilot Study): All groups

1. Poorly controlled hypertension, with blood pressure at study entry > 160 mmHg systolic or > 100 mmHg diastolic.
2. Current treatment with oral medication for diabetes.
3. Pregnant or nursing.
4. Participants unwilling or unable to undergo MR imaging, including patients with contra-indications to MRI, such as cardiac pacemakers or non-compatible intracranial vascular clips.
5. Participant size too large to fit in MR scanner.
6. Congestive heart failure with New York Heart Association (NYHA) status >= 2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients with diagnosed NASH or NAFLD, or adult healthy volunteers.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2020-07-22 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Optimal coil placement (Part 1) | 1 day
  Establishing suitable radiofrequency (RF) coils for individual applications and proper use of MRI techniques such as parallel imaging to achieve optimal image quality will be conducted during the participant's scan. There is no formal analytic plan for Part 1 of the study, which is focused on optimizing the image acquisition protocol.
Optimal pulse sequences (Part 1) | 1 day
  Establishing the pulse sequences for individual applications and proper use of MRI techniques such as parallel imaging to achieve optimal image quality will be conducted during the participant's scan. There is no formal analytic plan for Part 1 of the study, which is focused on optimizing the image acquisition protocol.
Optimal respiratory parameter (Part 1) | 1 day
  Establishing the magnitude of respiratory motion for individual applications and proper use of MRI techniques such as parallel imaging to achieve optimal image quality will be conducted during the participant's scan. There is no formal analytic plan for Part 1 of the study, which is focused on optimizing the image acquisition protocol.
Mean lactate/pyruvate conversion rate (kPL) (Part 1, Cohort B) | 1 day
  Mean lactate-to-pyruvate conversion will be calculated with 95% confidence intervals.
Signal-to-noise ratio (SNR) (Part 1, Cohort B) | 1 day
  SNR will be calculated..
Mean lactate-to-pyruvate ratio (Part 2) | 1 day
  The mean lactate-to-pyruvate ratio will be calculated for each of the diagnostic groups: (1) NAFL without steatohepatitis, (2) NASH, and (3) healthy volunteers.
Mean kPL(Part 2) | 1 day
  The mean kPL will be calculated for each of the diagnostic groups: (1) NAFL without steatohepatitis, (2) NASH, and (3) healthy volunteers.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Ohliger, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No